CLINICAL TRIAL: NCT01862692
Title: Web-based Parenting Intervention for Mothers of Infants At-Risk for Maltreatment
Brief Title: Web-based Parenting Intervention for Mothers of Infants At-Risk for Maltreatment (Baby-Net)
Acronym: Baby-Net
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01HD064870 (NIH)
Record Dates: First submitted 2013-05-01; First posted 2013-05-24 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Parenting

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Developmental Awareness Skils (Active Comparator)
  Interventions: Behavioral: Developmental Awareness Skills
- Baby-Net condition (Experimental)
  Interventions: Behavioral: Baby-Net

INTERVENTIONS:
Behavioral: Baby-Net — Parents randomized to the intervention condition will receive a computerized adaptation of the empirically supported PALS parenting program as well as a laptop and wireless Internet connection. In this study, we adapted original 10-session PALS program for computer administration and included a session on reading (Read to Me, Inc.; http://www.readtomeprogram.org/index.html), developed to be incorporated within the PALS program. Each session includes the following: (a) a presentation of concepts, behaviors, and examples, (b) check-in questions recorded to the data base for review by both parent and coach, (c) the creation of a 5 minute computer-collected video of mother-infant interactions for later review by coach and parent, (d) a summary of topics, (e) daily activities (homework), (f) feedback about the program recorded to the database and (g) a weekly telephone coach call to review mother-infant computer-administered video and session topics and skills.
  Arms: Baby-Net condition
Behavioral: Developmental Awareness Skills — Mothers in this condition will receive weekly phone contact with a coach as well as a laptop and wireless Internet connection. The laptop will contain a computer-based infant intervention program that is structurally similar to the Infant Program in terms of components (e.g., information pages, mother-infant video recording pages; coach contact pages), however weekly information will focus on their infants' development, with no direct maternal skills instruction. Mothers in this condition will receive the same number of contacts with the computer and coach as mothers in the InfantNet condition and will participate in weekly phone calls with a coach. During phone calls, parents will co-view weekly mother-infant video with their coach, with mothers having been instructed to play with their infant (with no prescribed tasks to perform) and the discussion will focus on general infant development.
  Arms: Developmental Awareness Skils

SUMMARY:
This innovative interactive Internet-based parent education intervention will help serve to promote the social emotional development and communication skills of infants to decrease the chances of child maltreatment in low-income, culturally diverse, families.

DETAILED DESCRIPTION:
Parents of infants living in poverty are at significantly elevated risk of a host of detrimental outcomes, including the development of child behavior problems, neglect and abuse of children, child learning problems and parental substance abuse. Research has found that early interventions to improve parenting practices were effective to ameliorate these outcomes. Yet, there exist major obstacles to the effective delivery of mental health services, particularly in rural areas. The need of rural families for mental health services is reaching crisis proportions due to the dearth of trained professionals. In addition, the meteoric rise of Internet use has created a new avenue for people to communicate and share ideas. These two trends are helping fuel the demand for mental health services and on-line support.

Internet programs can be interactive and provide social support from peers and professionals. Through the use of recent advances in multimedia technology and software as well as the rise of computer networking via the Internet, there now exists an opportunity to provide such monitoring of outcomes and remote contact for rural locations. Prior developmental R34 research ("Infant Net") successfully adapted and pilot tested an existing empirically proven parenting program, for delivery via the Internet, enhanced with weekly professional contact. This research provided 40 mothers of infants 3.5 to 7 months (at enrollment) with a computer, computer camera, Internet connection, and technical training/support for 6 months to evaluate the digital translation. Mother-infant dyads were randomized to Experimental or Computer/Control conditions. Results found significant change with infant-behavioral and positive trends were demonstrated in parenting behaviors. Mothers rated the both computer program and interaction with coaches to be very high. These encouraging developmental research results provide a very good empirical base for a fully powered randomized control trial to test effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18+ years old
* Child age 3.5-7.5 months
* Eligible for Early Head Start
* Understand spoken English or Spanish

Exclusion Criteria:

* History of severe drug use or psychopathology

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2011-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The Landry Parent-Child Interaction Scales (Parent Behavior) | 6 months post
  The Landry Scales are designed to assess naturalistic parent-child interaction. The parent scales of interest in the current study relative to maternal responsiveness include ratings of maternal positive affect, warmth, flexibility, and positive verbal content. Relative to maternal negative behavior, scales of interest include ratings of maternal physical intrusiveness as well as verbal and affective negativity.

SECONDARY OUTCOMES:
The Landry Parent-Child Interaction Scales (Infant Behavior) | 6 months (post)
  The Landry Parent-Child Interaction Scales, relative to directly observed maternal behavior, will also be used to assess infant functioning. Rating scales of interest in this regard are those assessing the infant behaviors of attention/arousal, warmth-seeking, and behavioral regulation. Ratings of infant behavior will be completed on the same mother-infant observational assessments as those used to assess maternal behavior at pre- and post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Ed G. Feil, Ph.D., Principal Investigator — Oregon Research Institute
Locations (2):
- United States (2):
  - University of Kansas Center for Research, Kansas City, Kansas
  - Oregon Research Institute, Eugene, Oregon